CLINICAL TRIAL: NCT01275014
Title: Corticosteroids as Additive in Arthrocentesis of the Temporomandibular Joint: Double Blind, Randomised Controlled Trial of Effectiveness.
Brief Title: Corticosteroids as Additive in Temporomandibular Joint (TMJ) Arthrocentesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: JJR Huddleston Slater, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMCG_KCHIR_01; 14439 (Other: Medical Ethical Committee University Medical Center)
Record Dates: First submitted 2010-11-29; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2010-11

CONDITIONS: Arthritis
Keywords: TMJ; corticosteroids; osteoarthritis; arthrocentesis; pain
MeSH Terms: conditions — Arthritis; Osteoarthritis; Pain | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Isotonic saline
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 1 ml of 20mg/ml solution was applied once, following the arthrocentesis procedure of the TMJ
  Arms: Dexamethasone
Drug: Isotonic saline — 1 ml of isotonic saline was applied once, following the arthrocentesis procedure of the TMJ
  Arms: Placebo

SUMMARY:
The aim is to compare the effectiveness of corticosteroid administration (dexamethasone) with a placebo (saline), following arthrocentesis of for the temporomandibular joint (TMJ). Twenty-eight participants with TMJ arthralgia, mainly related to osteoarthritis ae randomly assigned to two arms of a parallel double blind RCT. In both arms an arthrocentesis procedure is carried out, while a single dose intraarticular dexamethasone was delivered to participants in one arm. Saline was delivered in the other arm to serve as a control. Follow up visits were scheduled after 1, 3 and 24 weeks. During each visit TMJ pain (on a 100mm VAS) and joint stiffness (mouth opening in mm) are scored. Generalized estimating equations (GEE) are used for statistical analysis.

DETAILED DESCRIPTION:
The arthrocentesis procedure was performed under local anaesthesia and took place in a closed operation room under controlled conditions. After marking the points for insertion of the needles, a first 18 gauge injection needle was inserted into the upper intra-articular space of the TMJ. Correct positioning of the needle was determined by injecting and aspirating saline. Subsequently, a second 18 gauge needle was inserted into the upper joint space about 8-10 mm anterior of the first needle. Correct positioning of the second needle was confirmed by allowing injected saline to leave the joint through the first needle. After positioning of the needles, one needle was connected to a medical infusion system to passively allow isotonic saline of 37 degrees Celsius to enter the upper joint compartment. The other needle was connected to an outflow tube to allow the fluid to exit the joint. In about 15 minutes, approximately 300 ml saline passively flushed the joint. Thereafter, the inflow was stopped and the prepared syringe (see randomisation procedure) that contained either dexamethasone or saline was connected to the inflow needle. In this way, either 1 cc of dexamethasone or an equal amount of saline was washed through the joint in a blinded way. At the end of the procedure, the needles were removed from the joint, and after hemostasis by compression (if necessary) the skin overlying the TMJ was covered with a sterile band aid.

All patients were then instructed to avoid TMJ loading by following a soft diet for at least two weeks, then gradually advancing to more tough food. In addition, ibuprofen 600 mg 3dd was prescribed for the first 2-5 days to reduce any postoperative pain. All procedures were performed by one surgeon.

Follow up visits were scheduled after 1 (T1), 3 (T2) and 24 (T3) weeks.

ELIGIBILITY:
Inclusion Criteria:

Pain localized in one of the TMJs (TMJ arthralgia).

Exclusion Criteria:

* No significant relief of pain within 10 minutes after anaesthesia (injecting 0,1 ml articaine 40 mg/ml) of the TMJ
* Past history of open surgery in the affected joint
* Known polyarthritis (mostly rheumatoid arthritis)
* Age under 18 yrs
* Ankylosis of the TMJ
* Reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in TMJ pain at 24 weeks | 0 (T0), and at 1 (T1), 3 (T2) and 24 (T3) weeks.
  Change over 24 weeks from baseline for TMJ pain at rest and during mandibular movements. Measured by a 100 mm Visual Analogue Scale (VAS), limited by "no pain" and "worst pain imaginable".
Change from Baseline in Maximal interincisal opening at 24 weeks | T0, and at T1, T2 and T3.
  Change over 24 weeks from baseline maximal interincisal opening at rest and during mandibular movements . Measured in mm between the incisal edges of the center incisors.

SECONDARY OUTCOMES:
Change from baseline of mandibular function impairment at 24 weeks. | T0, T1, T2 and T3
  Change over 24 weeks from baseline for the MFIQ. The MFIQ is a questionnaire assessing, on a five point scale, discomfort while performing mandibular functions and during eating of food with different consistencies (range of 0 - 68).

CONTACTS AND LOCATIONS:
Overall Officials: James Huddleston Slater, PhD, Principal Investigator — University Medical Center
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Huddleston Slater JJ, Vos LM, Stroy LP, Stegenga B. Randomized trial on the effectiveness of dexamethasone in TMJ arthrocentesis. J Dent Res. 2012 Feb;91(2):173-8. doi: 10.1177/0022034511431260. Epub 2011 Dec 8. PMID 22157100